CLINICAL TRIAL: NCT06729580
Title: Risk-Targeted Behavioral Activation: a Novel Approach to the Management of Treatment-Resistant Depression.
Brief Title: Risk-Targeted Behavioural Activation for the Management of Treatment-Resistant Depression.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Responsible Party: Principal Investigator, Michael Sullivan, Principal investigator, McGill University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRC245719
Record Dates: First submitted 2024-09-30; First posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-09

CONDITIONS: Treatment Resistant Depression (TRD)
Keywords: treatment resistant depression; catastrophic thinking; perceived injustice; behavioural activation
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Behavioural Activation for Depression. (Experimental): All participants were enrolled in a 10-week standardized risk-targeted behavioural activation intervention.
  Interventions: Behavioral: Behavioural Activation

INTERVENTIONS:
Behavioral: Behavioural Activation — 10-week standardized behavioural activation program.

SUMMARY:
Depression is the leading cause of disability worldwide. Major Depressive Disorder (MDD) is the most common diagnosis made for individuals seeking treatment for depression. Although a wide range of treatments have been developed for the treatment of MDD, a significant proportion of patients fail to respond. This study examined the effectiveness of a 10-week behavioural activation intervention for individuals with treatment-resistant depression.

DETAILED DESCRIPTION:
Objective: The purpose of the present study was to examine the acceptability and impact of a standardized 10-week risk-targeted behavioral activation (RTBA) intervention as an augmentation strategy in the clinical management of treatment-resistant depression (TRD). Methods: The study sample consisted of 118 individuals with TRD, who were currently absent from work and referred to an occupational rehabilitation service. The RTBA intervention was a 10-week standardized program consisting of weekly visits with a trained clinician. The objectives of treatment included symptom reduction, resumption of important life activities (including return to work) and improvement in quality of life. Measures of depression, perceived injustice, and catastrophic thinking were completed pre-, mid- and post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of Major Depressive Disorder
* The date of diagnosis of MDD preceded referral by at least 12 months
* At least one previous prescription of an antidepressant failed to yield therapeutic response
* Currently taking an antidepressant
* A PHQ9 score in the moderate to severe range of depression at the time of enrolment

Exclusion Criteria:

- Participating in another psychotherapeutic intervention.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2022-01-05 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Depression symptom severity. | baseline/immediately after the intervention
  The Patient Health Questionnaire (PHQ9) was used to assess depressive symptom severity. PHQ-9 scores can range from 0 to 27 with higher scores indicating more severe depressive symptoms.

SECONDARY OUTCOMES:
Catastrophic thinking | baseline/immediately after the intervention.
  The Symptom Catastrophizing Scale (SCS) was used to assess catastrophic appraisals of depressive symptoms. Scores on the SCS range from 0 to 14 where higher scores reflect a higher degree of catastrophic thinking.
Perceived Injustice | baseline/immediately after the intervention.
  The Injustice Experience Questionnaire - Short Form (IEQ-SF) was used to assess injustice appraisals. Scores on the IEQ-SF range from 0 to 10 where higher scores reflect a greater sense of injustice.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Sullivan, PhD, Principal Investigator — McGill University; Heather Adams, BSW, Study Director — Dalhousie University
Locations (1):
- McGill University, Montreal, Quebec, Canada